CLINICAL TRIAL: NCT02812849
Title: Somatostatin Receptor Imaging in Cardiac Sarcoidosis
Status: Withdrawn | Type: Observational
Why Stopped: Logistic reasons
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Rasmus S. Ripa, MD, DMSc, Rigshospitalet, Denmark
Other Study IDs: 0001
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cardiac Sarcoidosis
MeSH Terms: interventions — copper dotatate CU-64

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Suspected cardiac sarcoidosis: Cu-64 DOTATATE PET/CT or PET/MRI
  Interventions: Drug: Cu-64 DOTATATE
- Known cardiac sarcoidosis: Cu-64 DOTATATE PET/CT or PET/MRI
  Interventions: Drug: Cu-64 DOTATATE
- Other inflammatory cardiac disease: Cu-64 DOTATATE PET/CT or PET/MRI
  Interventions: Drug: Cu-64 DOTATATE

INTERVENTIONS:
Drug: Cu-64 DOTATATE

SUMMARY:
The purpose of the trial is to determine the accuracy of Cu-64 labelled DOTATATE for diagnosing cardiac sarcoidosis using PET/CT or PET/MRI.

ELIGIBILITY:
Inclusion Criteria:

Group A: Suspected cardiac sarcoidosis Group B: Known cardiac sarcoidosis, clinical follow-up Group C: Myocarditis or dilated cardiomyopathy (Non-cardiac sarcoidosis)

Exclusion Criteria:

Infection Pregnancy Severe claustrophobia Weight >140 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or known cardiac sarcoidosis or with myocarditis/dilated cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2019-11 (Estimated); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Sensitivity to detect cardiac sarcoidosis | 1 day at PET/CT examination
Specificity to detect cardiac sarcoidosis | 1 day at PET/CT examination

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus S Ripa, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided